CLINICAL TRIAL: NCT07036406
Title: Comparing the Effectiveness of Traditional Semantic Feature Analysis (SFA) Versus SFA Plus Metacognitive Strategy Training (SFA+MST) for People With Acquired Aphasia
Brief Title: Comparing Traditional Semantic Feature Analysis (tSFA) and Semantic Feature Analysis + Metacognitive Strategy Training (SFA+MST)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Principal Investigator, Victoria Tilton-Bolowsky, Ph.D. CCC-SLP, Teachers College, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TeachersCCU
Record Dates: First submitted 2025-06-09; First posted 2025-06-25 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Aphasia; Aphasia Following Cerebral Infarction; Aphasia, Acquired; Aphasia, Rehabilitation; Aphasia, Anomic; Aphasia, Broca; Aphasia, Conduction; Aphasia, Expressive; Aphasia Non Fluent; Aphasia, Mixed
Keywords: Aphasia; Anomia; Stroke; Communication; Language
MeSH Terms: conditions — Aphasia; Anomia; Aphasia, Broca; Aphasia, Conduction; Stroke; Communication; Language

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Semantic Feature Analysis (Active Comparator): A portion of the study participants will participate in traditional Semantic Feature Analysis treatment, as described in Gravier, M. L., Dickey, M. W., Hula, W. D., Evans, W. S., Owens, R. L., Winans-Mitrik, R. L., & Doyle, P. J. (2018). What matters in semantic feature analysis: Practice-related predictors of treatment response in aphasia. American Journal of Speech-Language Pathology, 27(1S), 438-453. https://doi.org/10.1044/2017_AJSLP-16-0196. Briefly, this treatment involves naming pictures of objects, describing the objects' features (e.g., category membership, physical attributes, etc.), and creating sentences using the objects' names.
  Interventions: Behavioral: Semantic Feature Analysis (traditional)
- Semantic Feature Analysis + Metacognitive Strategy Training (Experimental): A portion of the study participants will participate in traditional Semantic Feature Analysis treatment, as described in Tilton-Bolowsky, V. E., Brock, L., Nunn, K., Evans, W. S., & Vallila-Rohter, S. (2023). Incorporating metacognitive strategy training into semantic treatment promotes restitutive and substitutive gains in naming: A single-subject investigation. American journal of speech-language pathology, 32(5), 1979-2020. https://doi.org/10.1044/2023_AJSLP-22-00230. Briefly, this treatment involves metacognitive teaching and practice, naming pictures of objects, describing the objects' features (e.g., category membership, physical attributes, etc), creating sentences using the objects' names, debriefing on overall performance, and discussing recent and future opportunities for strategy implementation in real life.
  Interventions: Behavioral: Semantic Feature Analysis + Metacognitive Strategy Training

INTERVENTIONS:
Behavioral: Semantic Feature Analysis (traditional) — This treatment involves naming pictures of objects, describing the objects' features (e.g., category membership, physical attributes, etc.), and creating sentences using the objects' names. It does not include direct metacognitive strategy training.
  Arms: Traditional Semantic Feature Analysis
Behavioral: Semantic Feature Analysis + Metacognitive Strategy Training — This treatment involves metacognitive teaching and practice, naming pictures of objects, describing the objects' features (e.g., category membership, physical attributes, etc), creating sentences using the objects' names, debriefing on overall performance, and discussing recent and future opportunities for strategy implementation in real life.
  Arms: Semantic Feature Analysis + Metacognitive Strategy Training

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of traditional Semantic Feature Analysis (SFA) treatment to a modified SFA protocol that includes Metacognitive Strategy Training (SFA+MST) for adults with acquired aphasia. The main questions it aims to answer are:

* What are the comparative outcomes in picture naming accuracy and strategy use during picture naming following 2 months of traditional SFA versus SFA + MST in adults with acquired aphasia?
* What are the comparative outcomes in percent of informative content and rate of informative content during spontaneous speech production following 2 months of traditional SFA versus SFA + MST in adults with acquired aphasia?

Researchers will compare outcomes between these two treatments to see if SFA+MST yields larger effects in picture naming and spontaneous speech outcomes than traditional SFA.

Participants will complete:

* 5-7 pre-treatment assessment sessions where they will be asked to name pictures, tell stories/describe pictures, answer questions, and complete questionnaires,
* 3 treatment sessions of SFA *OR* SFA+MST per week for 8 weeks, for a total of 24 sessions,
* 7 weekly probes (i.e., short, intermittent assessments throughout the treatment phase),
* 3 post-treatment assessment sessions immediately after treatment ends, where they will complete the same assessment tasks as they did pre-treatment (e.g., naming pictures, telling stories, etc.),
* 2 retention assessment sessions, one 30 days and the other 60 days following the final treatment session, where they will be asked to name pictures, tell stories/describe pictures, and describe what they learned during the study.

ELIGIBILITY:
Inclusion Criteria:

* Have aphasia due to a single acute event (e.g., left-hemisphere stroke, traumatic brain injury)
* Be at least six-months post aphasia-onset,
* Be a proficient English speaker,
* Have normal or corrected to normal hearing (i.e., hearing aids) and vision (i.e., eyeglasses),
* Have no history of neurodegenerative disease (e.g., dementia), severe motor speech disorder, significant mental illness, psychiatric disorder, drug/alcohol abuse, or neurological condition that could influence their cognitive, language, and memory systems

Exclusion Criteria:

* A history of neurodegenerative disease (e.g., dementia), severe motor speech disorder, significant mental illness, psychiatric disorder, drug/alcohol abuse, or neurological condition that could influence their cognitive, language, and memory systems,
* Children under the age of 18,
* Adults over the age of 89,
* Uncorrected hearing and vision.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Confrontation naming accuracy | Change from Baseline through study completion, an average of 6 months
  Participants will complete a 60-item confrontation naming assessment before, during, and after treatment. We will calculate the total number of items that participants name accurately across study phases.
Independent word-finding strategy use | Change from Baseline through study completion, an average of 6 months
  Using the 60-item confrontation naming assessment, we will evaluate instances in which participants independently use a specific word-finding strategy (describing or talking around the word) in instances where they cannot name items successfully, and calculate the proportions of incorrect responses with and without strategy use across study phases.

SECONDARY OUTCOMES:
Discourse informativeness | Change from Baseline through study completion, an average of 6 months
  Participants will describe picture scenes and tell stories. We will calculate the amount of informative content in their descriptions/stories using Content Information Unit (%CIU; Nicholas & Brookshire, 1993) analysis for descriptions/stories across study phases.
Discourse efficiency | Change from Baseline through study completion, an average of 6 months
  Participants will describe picture scenes and tell stories. We will calculate the rate of informative content in their descriptions/stories using Content Information Unit (CIU/minute; Nicholas & Brookshire, 1993) analysis for descriptions/stories across study phases.

OTHER OUTCOMES:
Explicit strategy knowledge | Change from Baseline through study completion, an average of 6 months
  Participants will be asked to identify what they can do in moments of word-finding difficulty and what types of information they can provide in those moments, across study phases. There are six types of information that will be discussed during the treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nicholas LE, Brookshire RH. A system for quantifying the informativeness and efficiency of the connected speech of adults with aphasia. J Speech Hear Res. 1993 Apr;36(2):338-50. doi: 10.1044/jshr.3602.338. PMID 8487525
- [Background] Gravier ML, Dickey MW, Hula WD, Evans WS, Owens RL, Winans-Mitrik RL, Doyle PJ. What Matters in Semantic Feature Analysis: Practice-Related Predictors of Treatment Response in Aphasia. Am J Speech Lang Pathol. 2018 Mar 1;27(1S):438-453. doi: 10.1044/2017_AJSLP-16-0196. PMID 29497754
- [Background] Tilton-Bolowsky VE, Brock L, Nunn K, Evans WS, Vallila-Rohter S. Incorporating Metacognitive Strategy Training Into Semantic Treatment Promotes Restitutive and Substitutive Gains in Naming: A Single-Subject Investigation. Am J Speech Lang Pathol. 2023 Sep 11;32(5):1979-2020. doi: 10.1044/2023_AJSLP-22-00230. Epub 2023 Jul 11. PMID 37433115